CLINICAL TRIAL: NCT01673347
Title: Allograft Knee Meniscal Transplantation in the Treatment of Osteoarthritis of the Metatarsophalangeal (MTP) Joint of the Great Toe
Brief Title: Allograft Transplantation in the Treatment of Osteoarthritis of the Metatarsophalangeal (MTP) Joint of the Great Toe
Acronym: MTP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paul Fortin, MD (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor-Investigator, Paul Fortin, MD, Orthopedic Surgeon, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-182; ISO 13485 (Other: MUSCULOSKELETAL TRANSPLANT FOUNDATION)
Record Dates: First submitted 2012-08-14; First posted 2012-08-28 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis
Keywords: allograft; great toe
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MENISCAL ALLOGRAFT (Experimental): The meniscal allograft is taken from the meniscal knee joint and implanted surgically in to the great toe.
  Interventions: Biological: Meniscal Allograft

INTERVENTIONS:
Biological: Meniscal Allograft — Meniscal allograft
  Other Names: Musculoskeletal Transplant Foundation; Meniscal transplant

SUMMARY:
Using the concept of an implant acting as a spacer and stabilizer, the proposed study will evaluate the use of allograft knee meniscus in the treatment of MTP joint osteoarthritis of the great toe.

DETAILED DESCRIPTION:
A variety of surgical procedures have been developed for the treatment of MTP joint osteoarthritis of the great toe. Using the concept of an implant acting as a spacer and stabilizer, the proposed study will evaluate the use of allograft knee meniscus in the treatment of MTP joint osteoarthritis of the great toe. Patients will be evaluated for pain and range of motion at 3-months, 6-months, 1-year, 2-years, 3-years, 4-years, and 5-years postoperatively or until allograft failure. Stability of the allograft will be evaluated by the surgeon at these time points per radiographic imaging.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic of stage 3 osteoarthritis of the great toe
* symptoms recalcitrant to nonoperative management as determined clinically by the principal investigator

Exclusion Criteria:

* diabetes mellitus
* kidney insufficiency
* oa in the adjacent joints
* malignancy with in the past 10 yrs
* minors (< 18 yrs of age)
* pregnant women and fetus
* mentally disabled or cognitively impaired individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PAUL FORTIN, MD, Principal Investigator — WILLIAM BEAUMONT HOSPITAL ROYAL OAK
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] COLE BJ, CARTER TR, RODEO SA,

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MENISCAL ALLOGRAFT
Started | 24
Completed | 17
Not Completed | 7
Not completed — failure of allograft | 7

BASELINE CHARACTERISTICS:
Arm/Group | MENISCAL ALLOGRAFT
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.27 (4.33)

OUTCOME MEASURES:

1. Primary Outcome: Allograft Stability
Description: Evaluation of the MTP joint space as determined by radiographic imaging. Count of participants maintaining adequate spacing and alignment as evaluated by the surgeon.
Time Frame: 5-years postoperative
Population: Study terminated prior to 5-year endpoint, no participants evaluated
Groups:
- MENISCAL ALLOGRAFT: The meniscal allograft is taken from the meniscal knee joint and implanted surgically in to the great toe for treatment of metatarsophalangeal (MTP) osteoarthritis.
Arm/Group | MENISCAL ALLOGRAFT
Number analyzed (Participants) | 0
Value | 0

2. Secondary Outcome: Pain
Description: Pain scored on Visual Analog Scale 0-10; 0 = no pain, 10 = worst pain
Time Frame: 3-months postoperative
Population: 17 participants available to analyze at 3 months due to early allograft failure in 7 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MENISCAL ALLOGRAFT
Number analyzed (Participants) | 17
units on a scale | 2.65 (2.13)

3. Secondary Outcome: Range of Motion Plantarflexion
Description: Range of Motion Plantarflexion
Time Frame: 3-months postoperative
Population: 17 participants available to analyze at 3 months due to early allograft failure in 7 participants
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | MENISCAL ALLOGRAFT
Number analyzed (Participants) | 17
degrees | 20 (8.13)

4. Secondary Outcome: Range of Motion Dorsiflexion
Description: Range of Motion Dorsiflexion
Time Frame: 3-months postoperative
Population: 17 participants available to analyze at 3 months due to early allograft failure in 7 participants
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | MENISCAL ALLOGRAFT
Number analyzed (Participants) | 17
degrees | 40 (15.86)

ADVERSE EVENTS:
Time Frame: 5 years postoperative
Arm/Group | MENISCAL ALLOGRAFT
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 7/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MENISCAL ALLOGRAFT (N=24)
Allograft failure (Musculoskeletal and connective tissue disorders) | 7 (7) — dissolution of allograft and obliteration of the MTP joint space

LIMITATIONS AND CAVEATS:
Allograft failure (dissolution) and obliteration of the MTP joint space found in 29% of subjects within 2 years of follow-up; therefore study was discontinued. No data collected for later time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No